CLINICAL TRIAL: NCT05815251
Title: Kiphoplasty With Porous Titanium Microspheres for Treatment of Vertebral Osteoporotic Compression Fractures: Perspective Study on Efficacy and Safety
Brief Title: Porous Titanium Microspheres in Kyphoplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unit of neurosurgery, Departement of Neurosciences, University of Torino (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Fabio Cofano, MD, Principal investigator, Researcher, Neurosurgeon, Unit of neurosurgery, Departement of Neurosciences, University of Torino
Other Study IDs: Microsphere001
Record Dates: First submitted 2023-02-24; First posted 2023-04-18 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Vertebral Fracture; Kyphoplasty
Keywords: osteoporotic fracture; vertebral augmentation; vertebral compression fracture
MeSH Terms: conditions — Spinal Fractures; Osteoporotic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sphereplast group: Patients with osteoporotic vertebral compression fractures identified as candidates for kyphoplasty treatment with porous trabecular titanium microspheres

SUMMARY:
Study is a prospective observational, performed in the context of normal clinical practice, of patients with osteoporotic vertebral compression fractures identified as candidates for kyphoplasty treatment with porous trabecular titanium microspheres (see whether to put commercial name and company). The study does not involve any interference with the patient's diagnostic-therapeutic course The objective of the study is the clinical-radiological evaluation of the efficacy of kyphoplasty treatment with trabecular porous titanium spheres in terms of pain control and reduction of kyphotic deformity following fracture. Further evaluation of the safety of the treatment in terms of absence of intraoperative adverse events and material-related toxicity.

DETAILED DESCRIPTION:
The study is purely observational, sponsored, and does not involve any change in the diagnostic, therapeutic, and follow-up course of patients selected on a clinical basis for kyphoplasty with porous titanium microspheres. involved but only an analysis and comparison of data during normal clinical-surgical activity. The study aims to evaluate, in a prospective-observational setting, the benefit of this treatment on pain control and prevention of deformity following fracture. Kyphoplasty with porous titanium spheres has already been used successfully and without obvious safety issues.

No additional radiologic exposures are planned over and above those in the normal courses of care and follow-up. No additional diagnostic investigations are planned. The study ensures data collection with full respect for privacy. There are no conflicts of interest for any of the board members.

The effectiveness of the therapy used is tested by considering the ODI, MRQ, VAS score expressed in numerical value before ("pre" condition) and after ("post" condition) kyphoplasty treatment as the observed quantity. The sample size is evaluated based on the primary objective of demonstrating a significant reduction in disability and pain after treatment in the range of 20%. With a significance of 0.05, a power of the test of 0.95, assuming to compare the two samples by t test for paired data the sample size can be in the order of 15 patients.

The evaluation of secondary end-points, which is not binding, will be carried out on similar sample numerosity.

All patients with the following requirements may be included in the observational study. The patient will be asked to give informed consent for inclusion in the study. Contextually, consent will be acquired for the processing of personal data in relation to the current privacy law. Consents must be acquired from the Investigating Surgeon performing the procedure in full respect of the Physician-Patient relationship. The informed consent will include acceptance of the follow-up period of at least 1 year with the possibility of telephone follow-up as well. The patient will also be given an information sheet regarding the purpose and type of the study and the expression of consent to participate. Attached is the informed consent form, patient information sheet and consent for personal data processing and privacy.

The procedure is performed under local anesthesia with the aid of possible sedation. Patient in prone position on radiolucent table with possibility of fluoroscopy in antero-posterior and latero-lateral projection. Biportal (bilateral) access with dedicated trokar to be placed in the anterior part of the fractured vertebral soma with convergent trajectory and transpeduncular access. Replacement of trokar with with larger cannula. Placement and dilatation of kyphoplasty balloon (15 ml volume) bilaterally. Introduction with dedicated instrument of porous titanium microspheres with possibility of using compactor to increase consistency of overall cast of material. Procedure performed with fluoroscopic control.

Data collection.

All data entered in the CRF data collection form must be collected for recruited patients:

* generality: age, sex, smoking habit, previous diagnosis of osteoporosis or new diagnosis of osteoporosis
* level and classification of fracture (AOSpine)
* operative data: date of surgery, type of access, number of spheres used, type of kyphoplasty pole, intraoperative adverse events, and technical difficulties
* clinical data: diagnosis, date of fracture, ODI, MRIQ, VAS back, days of postoperative hospital stay. For clinical and outcome assessment, point scales ODI score (Oswestry Disability Index) Roland-Morris Questionnaire, Back Pain Visual Analogue Scale (VAS) whose reliability is well reported in the literature (bibliographic entries) are used.
* Radiological data: segmental kyphosis, kyphosis of the fractured soma, possible progression of the fracture. Segmental kyphosis is calculated as Cobb angle, and changes (delta) pre-postoperative and at follow-up are reported.

Protection of privacy.

Data collection remains within the center promoting the research in the context of normal clinical activity and in compliance with current regulations. As reported, further consent to the processing of personal data is acquired. Radiological images will be obtained during the procedure and hospitalization will be archived regularly. Images performed externally in other hospitals or diagnostic centers will be acquired and stored, with the express consent of the patient, by the referring Investigating Surgeon. All images will eventually be used for scientific activities in a completely anonymous form.

All recruited patients should be followed, unless the patient explicitly withdraws consent, in follow-up for at least 1 year. the entire duration of the study initially planned to be 5 years. Follow-up evaluations will have to involve the acquisition of all data already indicated in section 4.4 to be entered in the data collection form (CRF-FU). The follow-up clinical evaluation will involve the acquisition of ODI, RMQ questionnaires in addition to VAS back at 1, 3 and 12 months.

Follow-up is the responsibility of the referring Investigating Surgeon in full respect of the Physician-Patient relationship and Privacy. A telephone evaluation may be performed on patients who are unavailable for outpatient evaluations or cannot be reached by administering ODI, RMQ and VAS back and interview.

Follow-up will also include the performance and acquisition of a lumbar spine X-ray performed in standing load at 1 month, 3 months and at 12 months as in the normal clinical course of patients undergoing percutaneous kyphoplasty procedures. Thus, patients are not subjected to additional examinations for participation in the study. Follow-up CT and MRI examinations will be performed eventually, as usual, only for supervening clinical reasons such as persistence of pain or appearance of new neurological deficits.

Participants in the study as investigators are all Surgeons with proven experience in spine surgery selected from within the medical team of the proposing center. Upon association of a Surgeon, a letter of intent in duplicate is required to be signed to emphasize the required commitment and the roles of the investigator.

Participating Investigating Surgeons may recruit patients in the context of their regular surgical practice. Recruitment should be prospective and the patient should be enrolled prior to kyphoplasty treatment in order to avoid selection bias related to the clinical outcome obtained.

ELIGIBILITY:
Inclusion Criteria:

* Presence of osteoporotic vertebral fracture occurred within the previous 6 weeks and documented by CT, MRI, or X-ray in relation to the diagnostic pathway the patient underwent
* Patients with fractures according to AO Spine-DGOU OF2, OF3 and OF4 classification are enrollable limited to cases in which soma height loss is less than 60% and in the absence of vertical split type pincer fracture.
* Diagnosis of osteoporosis preceding or concurrent with fracture occurrence, regardless of current therapy
* Favorable for inclusion in the study with signed informed consent, available for follow-up up to 1 year.
* Availability of adequate preoperative radiologic documentation: CT or MRI of the lumbar spine; RX required for evaluation of kyphosis.
* Availability of adequate and comprehensive clinical information including presence of ODI score, MRQ, VAS.

Exclusion Criteria:

* Presence of oncologic, metabolic, or endocrinologic diseases related to bone fragility
* Age < 55 years
* Previous treatment of arthrodesis, vertebroplasty, or percutaneous kyphoplasty for previous fractures
* Presence of neurological deficits in the lower limbs medullary or radicular prior to fracture occurrence
* Unavailability for follow-up for at least 1 year

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented presence of vertebral compression fracture/osteoporotic collapse. Osteoporosis is the most frequent bone disease with high incidence in the population over 55 years of age. The occurrence of vertebral compression fractures is very common in patients with osteoporosis either in association with minor trauma or as a spontaneous event.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disability index | 1 year
  Evaluation of the effectiveness of treatment on reducing disability secondary to the occurrence of osteoporotic compression fracture. The used scale is: Oswestry Disability Index (ODI) The effectiveness of the therapy used was tested by considering the ODI expressed (from 0 to 50) in numerical value before ("pre" condition) and after ("post" condition) kyphoplasty treatment as the observed quantity.
Patients with Pain improvement | 1 year
  Evaluation of the effectiveness of treatment on reducing pain after the treatment. The used scale is Back Pain Visual Analogue Scale (VAS) from 0 (no pain) to 10 (maximum pain).
  The effectiveness of the therapy used was tested by considering VAS scale expressed in numerical value before ("pre" condition) and after ("post" condition) kyphoplasty treatment as the observed quantity.

SECONDARY OUTCOMES:
Percentage of patients with side effects | 1 year
  Evaluation of treatment safety in terms of absence of side effects including neurological deficits, embolic phenomena, adverse reactions to the material
  , occurrence of surgical site infections, expressed in percentage (%) and in a binomial variable (less or more than 20%)
Rate of Kyphosis recovery | 3 months
  valuation of reduction by kyphoplasty treatment of kyphosis resulting from the fracture and deformation of the fractured vertebral body (segmental Cobb angle, degrees of kyphosis of the fractured soma)
Rate of patients with dislocation of the sphere | 1 year
  It t means the presence of a dislocation of the introduced material (the microspheres) outside the fractured vertebra, commonly understood as leakage.

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli studi di Torino, Turin, Italy

REFERENCES:
- [Background] Ravindra VM, Senglaub SS, Rattani A, Dewan MC, Hartl R, Bisson E, Park KB, Shrime MG. Degenerative Lumbar Spine Disease: Estimating Global Incidence and Worldwide Volume. Global Spine J. 2018 Dec;8(8):784-794. doi: 10.1177/2192568218770769. Epub 2018 Apr 24. PMID 30560029
- [Background] Martin BI, Mirza SK, Spina N, Spiker WR, Lawrence B, Brodke DS. Trends in Lumbar Fusion Procedure Rates and Associated Hospital Costs for Degenerative Spinal Diseases in the United States, 2004 to 2015. Spine (Phila Pa 1976). 2019 Mar 1;44(5):369-376. doi: 10.1097/BRS.0000000000002822. PMID 30074971
- [Background] Makino T, Kaito T, Fujiwara H, Honda H, Sakai Y, Takenaka S, Yoshikawa H, Yonenobu K. Risk Factors for Poor Patient-Reported Quality of Life Outcomes After Posterior Lumbar Interbody Fusion: An Analysis of 2-Year Follow-up. Spine (Phila Pa 1976). 2017 Oct 1;42(19):1502-1510. doi: 10.1097/BRS.0000000000002137. PMID 28248893
- [Background] Kaiser MG, Eck JC, Groff MW, Watters WC 3rd, Dailey AT, Resnick DK, Choudhri TF, Sharan A, Wang JC, Mummaneni PV, Dhall SS, Ghogawala Z. Guideline update for the performance of fusion procedures for degenerative disease of the lumbar spine. Part 1: introduction and methodology. J Neurosurg Spine. 2014 Jul;21(1):2-6. doi: 10.3171/2014.4.SPINE14257. PMID 24980578
- [Background] Costa F, Anania CD, Zileli M, Servadei F, Fornari M. Lumbar Spinal Stenosis: Introduction to the World Federation of Neurosurgical Societies (WFNS) Spine Committee Recommendations. World Neurosurg X. 2020 Mar 10;7:100075. doi: 10.1016/j.wnsx.2020.100075. eCollection 2020 Jul. PMID 32613188
- [Background] Eck JC, Sharan A, Ghogawala Z, Resnick DK, Watters WC 3rd, Mummaneni PV, Dailey AT, Choudhri TF, Groff MW, Wang JC, Dhall SS, Kaiser MG. Guideline update for the performance of fusion procedures for degenerative disease of the lumbar spine. Part 7: lumbar fusion for intractable low-back pain without stenosis or spondylolisthesis. J Neurosurg Spine. 2014 Jul;21(1):42-7. doi: 10.3171/2014.4.SPINE14270. PMID 24980584
- [Background] Wang JC, Dailey AT, Mummaneni PV, Ghogawala Z, Resnick DK, Watters WC 3rd, Groff MW, Choudhri TF, Eck JC, Sharan A, Dhall SS, Kaiser MG. Guideline update for the performance of fusion procedures for degenerative disease of the lumbar spine. Part 8: lumbar fusion for disc herniation and radiculopathy. J Neurosurg Spine. 2014 Jul;21(1):48-53. doi: 10.3171/2014.4.SPINE14271. PMID 24980585
- [Background] Resnick DK, Watters WC 3rd, Sharan A, Mummaneni PV, Dailey AT, Wang JC, Choudhri TF, Eck J, Ghogawala Z, Groff MW, Dhall SS, Kaiser MG. Guideline update for the performance of fusion procedures for degenerative disease of the lumbar spine. Part 9: lumbar fusion for stenosis with spondylolisthesis. J Neurosurg Spine. 2014 Jul;21(1):54-61. doi: 10.3171/2014.4.SPINE14274. PMID 24980586
- [Background] Resnick DK, Watters WC 3rd, Mummaneni PV, Dailey AT, Choudhri TF, Eck JC, Sharan A, Groff MW, Wang JC, Ghogawala Z, Dhall SS, Kaiser MG. Guideline update for the performance of fusion procedures for degenerative disease of the lumbar spine. Part 10: lumbar fusion for stenosis without spondylolisthesis. J Neurosurg Spine. 2014 Jul;21(1):62-6. doi: 10.3171/2014.4.SPINE14275. PMID 24980587
- [Background] Groff MW, Dailey AT, Ghogawala Z, Resnick DK, Watters WC 3rd, Mummaneni PV, Choudhri TF, Eck JC, Sharan A, Wang JC, Dhall SS, Kaiser MG. Guideline update for the performance of fusion procedures for degenerative disease of the lumbar spine. Part 12: pedicle screw fixation as an adjunct to posterolateral fusion. J Neurosurg Spine. 2014 Jul;21(1):75-8. doi: 10.3171/2014.4.SPINE14277. PMID 24980589